CLINICAL TRIAL: NCT01827384
Title: Molecular Profiling-Based Assignment of Cancer Therapy for Patients With Advanced Solid Tumors
Brief Title: MPACT Study to Compare Effects of Targeted Drugs on Tumor Gene Variations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-01588; NCI-2013-01588 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MPACT; 130105; P121047; 9149 (Other: National Cancer Institute LAO); 9149 (Other: CTEP); ZIABC011078 (NIH)
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Results first posted 2022-05-10 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Advanced Malignant Solid Neoplasm
MeSH Terms: interventions — adavosertib; Carboplatin; Everolimus; Temozolomide; trametinib; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Regimen I (veliparib, temozolomide) (Experimental): Patients receive veliparib by mouth (PO) twice a day (BID) on days 1-7 and temozolomide PO every day (QD) on days 1-5. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Temozolomide; Drug: Veliparib
- Regimen II (adavosertib, carboplatin) (Experimental): Patients receive adavosertib by mouth (PO) twice a day (BID) for 5 doses starting on day 1 and carboplatin intravenous (IV) over 30-60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Adavosertib; Drug: Carboplatin
- Regimen III (everolimus) (Experimental): Patients receive everolimus by mouth (PO) every day (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Everolimus
- Regimen IV (trametinib) (Experimental): Patients receive trametinib by mouth (PO) every day (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Trametinib

INTERVENTIONS:
Drug: Adavosertib — Given by mouth (PO)
  Other Names: AZD-1775; AZD1775; MK-1775; MK1775
  Arms: Regimen II (adavosertib, carboplatin)
Drug: Carboplatin — Given intravenous (IV)
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Regimen II (adavosertib, carboplatin)
Drug: Everolimus — Given by mouth (PO)
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD001; Votubia; Zortress
  Arms: Regimen III (everolimus)
Drug: Temozolomide — Given by mouth (PO)
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ
  Arms: Regimen I (veliparib, temozolomide)
Drug: Trametinib — Given by mouth (PO)
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212
  Arms: Regimen IV (trametinib)
Drug: Veliparib — Given by mouth (PO)
  Other Names: ABT-888; PARP-1 inhibitor ABT-888
  Arms: Regimen I (veliparib, temozolomide)

SUMMARY:
This phase II trial studies molecular profiling-based assignment of cancer therapy (MPACT) in treating patients with solid tumors that have spread to other places in the body and usually cannot be cured or controlled with treatment (advanced). Adavosertib, everolimus, and trametinib are drugs that each target a specific variation in tumors by blocking different proteins needed for cell growth. Veliparib blocks an enzyme that helps repair deoxyribonucleic acid (DNA) damaged by chemotherapy, which may help chemotherapy drugs work better. It is not yet known whether testing patients for variations in their tumor and assigning treatment targeting the variation is more effective than standard non-targeted therapy in treating advanced solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers.

OUTLINE: Patients are assigned to 1 of 4 treatment regimens corresponding to one of their mutation/amplification categories.

REGIMEN I: Patients receive veliparib orally (PO) twice daily (BID) on days 1-7 and temozolomide PO once daily (QD) on days 1-5. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

REGIMEN II: Patients receive adavosertib PO BID for 5 doses starting on day 1 and carboplatin intravenously (IV) over 30-60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. (No longer an active study drug as of March 2018)

REGIMEN III: Patients receive everolimus PO every day (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. (No longer an active study drug as of March 2018)

REGIMEN IV: Patients receive trametinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. (No longer an active study drug as of March 2018)

After completion of study treatment, patients are followed up for 30 days. Patients with unacceptable toxicities that have not resolved by day 30 are followed up biweekly until stabilization or resolution.

ELIGIBILITY:
Inclusion Criteria:

* TUMOR BIOPSY SEQUENCING: Patients with histologically documented solid tumors whose disease has progressed following at least one line of standard therapy and/or no standard of treatment exists that has been shown to prolong survival
* TUMOR BIOPSY SEQUENCING: Patient must have tumor amenable to percutaneous or excisional skin biopsy and be willing to undergo a tumor biopsy or biopsy samples (formalin-fixed paraffin-embedded [FFPE] blocks) collected on another study or from a procedure performed due to medical necessity may be acceptable if collected within 6 months prior to registration on molecular profiling-based assignment of cancer therapy (MPACT) and providing that the patient has not received any investigational or targeted treatment since that time, or a report from a Molecular Analysis for Therapy Choice (MATCH) study designated Clinical Laboratory Improvement Act (CLIA) laboratory that a patient has a variant in the genes of interest
* TUMOR BIOPSY SEQUENCING: Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan
* TUMOR BIOPSY SEQUENCING: Patients with bone metastases or hypercalcemia on intravenous bisphosphonate treatment, denosumab, or similar agents are eligible to participate and may continue this treatment; patients with prostate cancer may continue luteinizing hormone-releasing hormone (LHRH) agonists or antagonists
* TUMOR BIOPSY SEQUENCING: Karnofsky performance status >= 70%
* TUMOR BIOPSY SEQUENCING: Life expectancy > 3 months
* TUMOR BIOPSY SEQUENCING: Absolute neutrophil count >= 1,000/uL (mcL)
* TUMOR BIOPSY SEQUENCING: Platelets >= 100,000/uL (mcL)
* TUMOR BIOPSY SEQUENCING: Total bilirubin < 1.5 x institutional upper limit of normal
* TUMOR BIOPSY SEQUENCING: Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional upper limit of normal
* TUMOR BIOPSY SEQUENCING: Creatinine < 1.5 x institutional upper limit of normal OR creatinine clearance >= 60 mL/min for patients with creatinine levels >= 1.5 x institutional upper limit of normal
* TUMOR BIOPSY SEQUENCING: The effects of these targeted agents on the developing human fetus are unknown or anticipated to cause fetal harm based on their mechanism of action; for this reason, women of childbearing potential and men must agree to use highly effective contraception prior to study entry, for the duration of study participation, and for 3 months after completion of study; because there may be a risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued while the patient is on this trial and for 30 days following last dose of study drug
* TUMOR BIOPSY SEQUENCING: Patients with history of central nervous system (CNS) metastases who have received treatment and who either have not had seizures or have been on stable doses of anti-seizure medicine and had no seizures for 4 weeks will be eligible; enzyme-inducing anticonvulsants are contraindicated
* TUMOR BIOPSY SEQUENCING: Ability to understand and the willingness to sign a written informed consent document (subjects with impaired decision-making capacity are not eligible)
* TREATMENT: Patient must have predefined targeted mutation in tumor biopsy
* TREATMENT: Patients with histologically documented solid tumors whose disease has progressed following at least one line of standard therapy or for which no standard therapy exists that has been shown to prolong survival
* TREATMENT: Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* TREATMENT: Any prior therapy, radiotherapy, or major surgery must have been completed >= 3 weeks (> 6 weeks for nitrosoureas or mitomycin C) or 5 half-lives of the agent (whichever is shorter) prior to enrollment on protocol, and the participant must have recovered to eligibility levels from prior toxicity; radiofrequency ablation (RFA) of localized lesions should have been performed >= 2 weeks prior to treatment
* TREATMENT: Patients with bone metastases or hypercalcemia on intravenous bisphosphonate treatment, denosumab, or similar agents are eligible to participate and may continue this treatment; patients with prostate cancer may continue LHRH agonists or antagonists
* TREATMENT: Karnofsky performance status >= 70%
* TREATMENT: Absolute neutrophil count >= 1,000/uL (mcL)
* TREATMENT: Platelets >= 100,000/uL (mcL)
* TREATMENT: Total bilirubin < 1.5 x institutional upper limit of normal
* TREATMENT: AST (SGOT)/ALT (SGPT) =< 3 x institutional upper limit of normal
* TREATMENT: Creatinine < 1.5 x institutional upper limit of normal OR creatinine clearance >= 60 mL/min for patients with creatinine levels >= 1.5 x institutional upper limit of normal
* TREATMENT: Life expectancy > 3 months
* TREATMENT: The effects of these targeted agents on the developing human fetus are unknown or anticipated to cause fetal harm based on their mechanism of action; for this reason, women of childbearing potential and men must agree to use highly effective contraception (see list below) prior to study entry, for the duration of study participation, and for 3 months after completion of study;

  * Total abstinence: When this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
  * Sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment
  * In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate); (for female subjects on the study, the vasectomized male partner should be the sole partner for that subject); use of a combination of any two of the following:
  * Use of oral, injected, implanted or other hormonal methods of contraception
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
  * In case of use of oral contraception, women should have been stable on the oral agent before taking study treatment
  * Sexually active males must use a condom during intercourse
* TREATMENT: Because there may be a risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued while the patient is on this trial and for 30 days following last dose of study drug
* TREATMENT: Patients with ovarian cancer or metastatic breast cancer and breast cancer gene (BRCA) mutations must have received approved poly (ADP-ribose) polymerase (PARP) inhibitor therapy; these patients are eligible for the veliparib plus temozolomide arm unless the PARP inhibitor was administered with temozolomide
* TREATMENT: Patients with a history of seizures are not eligible to receive veliparib
* TREATMENT: Patients who have had prior treatment with any PARP inhibitor in combination with temozolomide are not eligible to receive treatment with veliparib on this study; patients who have received prior temozolomide or PARP inhibitor with or without other chemotherapy/targeted agent should not be excluded
* TREATMENT: Patients must have >= 10.0 g/dL hemoglobin (Hb) and no blood transfusion in the past 28 days to receive veliparib

Exclusion Criteria:

* TUMOR BIOPSY SEQUENCING: Women who are pregnant or breastfeeding
* TUMOR BIOPSY SEQUENCING: Patients who are receiving any other investigational agents; patients on other trials will be eligible as long as they are no longer receiving study treatment
* TUMOR BIOPSY SEQUENCING: Patients with uncontrolled intercurrent illness including, but not limited to psychiatric illness/social situations that would limit compliance with study requirements, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, myocardial infarction in the past 6 months, invasive fungal infections, or active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and active and chronic hepatitis (i.e., quantifiable hepatitis B virus [HBV]-DNA and/or positive hepatitis B surface antigen [HbsAg], quantifiable hepatitis C virus [HCV]-ribonucleic acid [RNA]) are not eligible to participate; testing for hepatitis B or other infections for eligibility will be performed only if clinically indicated
* TUMOR BIOPSY SEQUENCING: Patients with gastrointestinal conditions that might predispose for drug intolerability or poor drug absorption (e.g., inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, malabsorption syndrome, and active peptic ulcer disease) are excluded; subjects with Crohn's disease or a partial or complete small bowel obstruction are also excluded, as are any patients who cannot swallow tablets or capsules whole; tablets or capsules must not be crushed or chewed; nasogastric or gastrostomy tube (G-tube) administration is not allowed
* TUMOR BIOPSY SEQUENCING: Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic (PK) interactions
* TUMOR BIOPSY SEQUENCING: Patients who require use of coumarin-derivative anticoagulants such as warfarin are excluded; low molecular weight heparin is permitted for prophylactic or therapeutic use
* TUMOR BIOPSY SEQUENCING: Patients who have previously been treated with the combination of temozolomide plus a PARP inhibitor should not be considered eligible for a biopsy given that these patients would not be eligible for the active veliparib plus temozolomide arm
* TREATMENT: Women who are pregnant or breastfeeding
* TREATMENT: Patients who are receiving any other investigational agents; patients on other trials will be eligible as long as they are no longer receiving study treatment
* TREATMENT: Patients with active brain metastases or carcinomatous meningitis are excluded from this clinical trial; patients who have a history of seizures are not eligible to receive veliparib
* TREATMENT: Patients with uncontrolled intercurrent illness including, but not limited to psychiatric illness/social situations that would limit compliance with study requirements, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, myocardial infarction in the past 6 months, invasive fungal infections, or active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and active and chronic hepatitis (i.e., quantifiable hepatitis B virus (HBV)-DNA and/or positive hepatitis B surface antibody (HbsAg), quantifiable hepatitis C virus (HCV)-RNA) are not eligible to participate; testing for hepatitis B or other infections for eligibility will be performed only if clinically indicated
* TREATMENT: Patients with gastrointestinal conditions that might predispose for drug intolerability or poor drug absorption (e.g., inability to take oral medication or a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, malabsorption syndrome, and active peptic ulcer disease) are excluded; subjects with Crohn's disease or a partial or complete small bowel obstruction are also excluded, as are any patients who cannot swallow tablets or capsules whole; tablets or capsules must not be crushed or chewed; nasogastric or G-tube administration is not allowed
* TREATMENT: HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for PK interactions
* TREATMENT: Eligibility of subjects receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics (i.e., cytochrome P450, family 3, subfamily A, polypeptide 4 [CYP450], P-glycoprotein [PgP]) of any of the study drugs will be determined following review of their cases by the principal investigator (PI); patients on strong and moderate cytochrome P450 system inducers or inhibitors are ineligible; every effort would be made to switch patients off medications that are known substrates of CYP450; if it is medically important for the patient to remain on such medications, these patients can still be eligible to participate based on PI discretion
* TREATMENT: Patients who require use of coumarin-derivative anticoagulants such as warfarin are excluded; low molecular weight heparin is permitted for prophylactic or therapeutic use
* TREATMENT: Patients who have a history of another primary malignancy, with the exceptions of: non-melanoma skin cancer, and carcinoma in situ of the cervix, uteri, or breast from which the patient has been disease free for > 3 years
* TREATMENT: Patients with treatment-related acute myeloid leukemia (AML) (t-AML)/myelodysplastic syndrome (MDS), or with features suggestive of AML/MDS, or who have had prior allogeneic bone marrow transplant or double umbilical cord blood transplantation, should not receive veliparib due to reports of MDS and leukemia secondary to oncology therapy on Cancer Therapy Evaluation Program (CTEP)-sponsored studies utilizing veliparib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2014-01-07 (Actual); Primary Completion 2021-06-19 (Actual); Study Completion 2021-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A P Chen, Principal Investigator — National Cancer Institute LAO
Locations (8):
- United States (8):
  - University of Colorado Hospital, Aurora, Colorado
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lih CJ, Sims DJ, Harrington RD, Polley EC, Zhao Y, Mehaffey MG, Forbes TD, Das B, Walsh WD, Datta V, Harper KN, Bouk CH, Rubinstein LV, Simon RM, Conley BA, Chen AP, Kummar S, Doroshow JH, Williams PM. Analytical Validation and Application of a Targeted Next-Generation Sequencing Mutation-Detection Assay for Use in Treatment Assignment in the NCI-MPACT Trial. J Mol Diagn. 2016 Jan;18(1):51-67. doi: 10.1016/j.jmoldx.2015.07.006. Epub 2015 Nov 18. PMID 26602013

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Assignment Code 1 (TAC1): TAC1: Veliparib (ABT-888) 40mg by mouth (PO) twice a day (BID) on days 1-7; Temozolomide 150 mg/m^2 PO every day (QD) on days 1-5
- TAC1 -> TAC4: TAC1: Veliparib (ABT-888) 40mg by mouth (PO) twice a day (BID) on days 1-7; Temozolomide 150 mg/m^2 PO every day (QD) on days 1-5 TAC4: Adavosertib (MK-1775) 225 mg by mouth (PO) twice a day (BID) x 5 doses on days 1-3; Carboplatin area under the concentration (AUC) 5 intravenous (IV) over 30 min on day 1
- TAC2: TAC2: Everolimus 10 mg by mouth (PO) every day (QD)
- TAC2 -> TAC1: TAC2: Everolimus 10 mg by mouth (PO) every day (QD) TAC1: Veliparib (ABT-888) 40mg by mouth (PO) twice a day (BID) on days 1-7; Temozolomide 150 mg/m^2 PO every day (QD) on days 1-5
- TAC2 -> TAC3: TAC2: Everolimus 10 mg by mouth (PO) every day (QD) TAC3: Trametinib 2mg by mouth (PO) every day (QD)
- TAC3: TAC3: Trametinib 2mg by mouth (PO) every day (QD)
- TAC3 -> TAC1: TAC3: Trametinib 2mg by mouth (PO) every day (QD) TAC1: Veliparib (ABT-888) 40mg by mouth (PO) twice a day (BID) on days 1-7; Temozolomide 150 mg/m^2 PO every day (QD) on days 1-5
- TAC3 -> TAC1 -> TAC4: TAC3: Trametinib 2mg by mouth (PO) every day (QD) TAC1: Veliparib (ABT-888) 40mg by mouth (PO) twice a day (BID) on days 1-7; Temozolomide 150 mg/m^2 PO every day (QD) on days 1-5 TAC4: Adavosertib (MK-1775) 225 mg by mouth (PO) twice a day (BID) x 5 doses on days 1-3; Carboplatin area under the concentration (AUC) 5 intravenous (IV) over 30 min on day 1
- TAC3 -> TAC4: TAC3: Trametinib 2mg by mouth (PO) every day (QD) TAC4: Adavosertib (MK-1775) 225 mg by mouth (PO) twice a day (BID) x 5 doses on days 1-3; Carboplatin area under the concentration (AUC) 5 intravenous (IV) over 30 min on day 1
- TAC4: TAC4: Adavosertib (MK-1775) 225 mg by mouth (PO) twice a day (BID) x 5 doses on days 1-3; Carboplatin area under the concentration (AUC) 5 intravenous (IV) over 30 min on day 1
- TAC4 -> TAC1: TAC4: Adavosertib (MK-1775) 225 mg by mouth (PO) twice a day (BID) x 5 doses on days 1-3; Carboplatin area under the concentration (AUC) 5 intravenous (IV) over 30 min on day 1 TAC1: Veliparib (ABT-888) 40mg by mouth (PO) twice a day (BID) on days 1-7; Temozolomide 150 mg/m^2 PO every day (QD) on days 1-5
- TAC4 -> TAC2: TAC4: Adavosertib (MK-1775) 225 mg by mouth (PO) twice a day (BID) x 5 doses on days 1-3; Carboplatin area under the concentration (AUC) 5 intravenous (IV) over 30 min on day 1 TAC2: Everolimus 10 mg by mouth (PO) every day (QD)
- TAC4 -> TAC3: TAC4: Adavosertib (MK-1775) 225 mg by mouth (PO) twice a day (BID) x 5 doses on days 1-3; Carboplatin area under the concentration (AUC) 5 intravenous (IV) over 30 min on day 1 TAC3: Trametinib 2mg by mouth (PO) every day (QD)
- Participants Enrolled But Not Treated: Participants who signed consent and were enrolled but not treated.
Period: Overall Study
Arm/Group | Treatment Assignment Code 1 (TAC1) | TAC1 -> TAC4 | TAC2 | TAC2 -> TAC1 | TAC2 -> TAC3 | TAC3 | TAC3 -> TAC1 | TAC3 -> TAC1 -> TAC4 | TAC3 -> TAC4 | TAC4 | TAC4 -> TAC1 | TAC4 -> TAC2 | TAC4 -> TAC3 | Participants Enrolled But Not Treated
Started | 13 | 1 | 9 | 1 | 1 | 22 | 2 | 1 | 2 | 15 | 7 | 1 | 2 | 131
Completed | 13 | 1 | 9 | 1 | 1 | 22 | 2 | 1 | 2 | 15 | 7 | 1 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 131
Not completed — Switched to alternative treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Disease progression before treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Ineligible | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19
Not completed — Participant died before treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Insufficient tumor cells | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13
Not completed — No actionable mutation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 73
Not completed — Participant declined to participate (before treatment started) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15

BASELINE CHARACTERISTICS:
Population: Enrollment data was captured for 131 participants who signed consent and were enrolled but not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Assignment Code 1 (TAC1) | TAC1 -> TAC4 | TAC2 | TAC2 -> TAC1 | TAC2 -> TAC3 | TAC3 | TAC3 -> TAC1 | TAC3 -> TAC1 -> TAC4 | TAC3 -> TAC4 | TAC4 | TAC4 -> TAC1 | TAC4 -> TAC2 | TAC4 -> TAC3 | Participants Enrolled But Not Treated | Total
Number analyzed (Participants) | 13 | 1 | 9 | 1 | 1 | 22 | 2 | 1 | 2 | 15 | 7 | 1 | 2 | 131 | 208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 1 | 6 | 1 | 1 | 13 | 2 | 1 | 2 | 11 | 3 | 1 | 2 | 89 | 139
  >=65 years | 7 | 0 | 3 | 0 | 0 | 9 | 0 | 0 | 0 | 4 | 4 | 0 | 0 | 42 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (15.15) | 59 (0) | 54 (15.15) | 59.1 (0) | 59 (0) | 58 (12.22) | 54 (9.9) | 45 (0) | 55.95 (7) | 59 (10.54) | 63.2 (13.72) | 39 (0) | 61.65 (4.03) | 58 (11.53) | 57.75 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 0 | 6 | 1 | 1 | 12 | 1 | 0 | 2 | 13 | 3 | 1 | 0 | 67 | 116
  Male | 4 | 1 | 3 | 0 | 0 | 10 | 1 | 1 | 0 | 2 | 4 | 0 | 2 | 64 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 11 | 15
  Not Hispanic or Latino | 13 | 1 | 8 | 1 | 1 | 19 | 2 | 1 | 2 | 14 | 7 | 1 | 2 | 117 | 189
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 9 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 19 | 28
  White | 11 | 1 | 8 | 1 | 1 | 15 | 2 | 1 | 2 | 9 | 5 | 1 | 2 | 95 | 154
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 13 | 1 | 9 | 1 | 1 | 22 | 2 | 1 | 2 | 15 | 7 | 1 | 2 | 131 | 208
Karnofsky Performance Status [Count of Participants; unit: Participants] — Karnofsky Performance Status 100 = Normal, no complaints, no evidence of disease. 90 = Able to carry on normal activity; minor signs or symptoms of disease. 80 = Normal activity with effort; some signs or symptoms of disease. 70 = Cares for self, unable to carry on normal activity or to do active work. 100 is a better outcome than 70.
  Participants
    100 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 6 | 11
    90 | 8 | 1 | 2 | 1 | 1 | 14 | 2 | 0 | 0 | 8 | 4 | 1 | 1 | 76 | 119
    80 | 3 | 0 | 6 | 0 | 0 | 6 | 0 | 1 | 1 | 6 | 2 | 0 | 1 | 41 | 67
    70 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 11
Participants with an Actionable Mutation of Interest (aMOI) in a Targeted Pathway [Count of Participants; unit: Participants] — Reported for all participants with an aMOI (i.e. mutations of interest) detected. Participants with an aMOI in more than one pathway are counted here by mutation with highest frequency. Therefore, rows are mutually exclusive; a participant cannot be counted in more than 1 row.
  PI3K - phosphoinositide 3-kinase RAF - rapidly accelerated fibrosarcoma RAS - rat sarcoma MEK - mitogen-activated protein kinase/extracellular signal-regulated kinase (ERK) No aMOI detected - Biopsy either was not collected, could not be analyzed, or did not have an aMOI detected.
  Participants
    Deoxyribonucleic acid (DNA) repair | 9 | 1 | 5 | 0 | 0 | 4 | 1 | 1 | 1 | 11 | 7 | 0 | 1 | 21 | 62
    P13K | 1 | 0 | 4 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 4 | 15
    RAS/RAF/MEK | 3 | 0 | 0 | 1 | 0 | 17 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 13 | 38
    No aMOI detected | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 93 | 93

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Objective Response
Description: ORR is the proportion of participants with a complete response (CR) or partial response (PR) per the Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response is disappearance of all tumors. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to 30 days after completion of study treatment, up to 75 months
Population: Participants enrolled but not treated were not applicable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Assignment Code 1 (TAC1) | TAC1 -> TAC4 | TAC2 | TAC2 -> TAC1 | TAC2 -> TAC3 | TAC3 | TAC3 -> TAC1 | TAC3 -> TAC1 -> TAC4 | TAC3 -> TAC4 | TAC4 | TAC4 -> TAC1 | TAC4 -> TAC2 | TAC4 -> TAC3
Number analyzed (Participants) | 13 | 1 | 9 | 1 | 1 | 22 | 2 | 1 | 2 | 15 | 7 | 1 | 2
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Proportion of Participants With 4 Month Progression-free Survival (PFS)
Description: Time from random assignment to progression or death from any cause (whichever comes first). Progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST). Progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. And the appearance of one or more new lesions is also considered progressions.
Time Frame: 4 months
Population: Participants enrolled but not treated were not applicable for this outcome measure.
Measure: Number; unit: proportion of participants
Arm/Group | Treatment Assignment Code 1 (TAC1) | TAC1 -> TAC4 | TAC2 | TAC2 -> TAC1 | TAC2 -> TAC3 | TAC3 | TAC3 -> TAC1 | TAC3 -> TAC1 -> TAC4 | TAC3 -> TAC4 | TAC4 | TAC4 -> TAC1 | TAC4 -> TAC2 | TAC4 -> TAC3
Number analyzed (Participants) | 13 | 1 | 9 | 1 | 1 | 22 | 2 | 1 | 2 | 15 | 7 | 1 | 2
proportion of participants | 0.23 | 0.00 | 0.22 | 0.00 | 1.00 | 0.41 | 0.50 | 0.00 | 0.00 | 0.13 | 0.29 | 0.00 | 0.00

3. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approx. 73months (m) & 21day (d); 4m & 11d; 61m & 8d; 4m & 11d; 10m & 11d; 72m & 29d; 13m & 11d; 6m & 13d; 29m & 18d; 48m & 25d; 49m & 5d; 4m &7d; 15m & 5d; and 75m &13d, for each group respectively.
Population: Adverse events were collected for participants that were enrolled but not treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Assignment Code 1 (TAC1) | TAC1 -> TAC4 | TAC2 | TAC2 -> TAC1 | TAC2 -> TAC3 | TAC3 | TAC3 -> TAC1 | TAC3 -> TAC1 -> TAC4 | TAC3 -> TAC4 | TAC4 | TAC4 -> TAC1 | TAC4 -> TAC2 | TAC4 -> TAC3 | Participants Enrolled But Not Treated
Number analyzed (Participants) | 13 | 1 | 9 | 1 | 1 | 22 | 2 | 1 | 2 | 15 | 7 | 1 | 2 | 131
Participants | 13 | 1 | 9 | 1 | 1 | 22 | 2 | 1 | 2 | 15 | 7 | 1 | 2 | 2

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 73months (m) & 21day (d); 4m & 11d; 61m & 8d; 4m & 11d; 10m & 11d; 72m & 29d; 13m & 11d; 6m & 13d; 29m & 18d; 48m & 25d; 49m & 5d; 4m &7d; 15m & 5d; and 75m &13d, for each group respectively.
Arm/Group | Treatment Assignment Code 1 (TAC1) | TAC1 -> TAC4 | TAC2 | TAC2 -> TAC1 | TAC2 -> TAC3 | TAC3 | TAC3 -> TAC1 | TAC3 -> TAC1 -> TAC4 | TAC3 -> TAC4 | TAC4 | TAC4 -> TAC1 | TAC4 -> TAC2 | TAC4 -> TAC3 | Participants Enrolled But Not Treated
All-Cause Mortality (participants affected / at risk) | 1/13 | 0/1 | 3/9 | 0/1 | 0/1 | 1/22 | 0/2 | 0/1 | 0/2 | 1/15 | 1/7 | 0/1 | 0/2 | 5/131
Serious Adverse Events (participants affected / at risk) | 5/13 | 0/1 | 4/9 | 1/1 | 0/1 | 11/22 | 1/2 | 1/1 | 1/2 | 10/15 | 4/7 | 1/1 | 2/2 | 10/131
Other Adverse Events (participants affected / at risk) | 13/13 | 1/1 | 9/9 | 1/1 | 1/1 | 22/22 | 2/2 | 1/1 | 2/2 | 15/15 | 7/7 | 1/1 | 2/2 | 2/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Assignment Code 1 (TAC1) (N=13) | TAC1 -> TAC4 (N=1) | TAC2 (N=9) | TAC2 -> TAC1 (N=1) | TAC2 -> TAC3 (N=1) | TAC3 (N=22) | TAC3 -> TAC1 (N=2) | TAC3 -> TAC1 -> TAC4 (N=1) | TAC3 -> TAC4 (N=2) | TAC4 (N=15) | TAC4 -> TAC1 (N=7) | TAC4 -> TAC2 (N=1) | TAC4 -> TAC3 (N=2) | Participants Enrolled But Not Treated (N=131)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 1 (1) | 1 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, CNS Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, ureter obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Assignment Code 1 (TAC1) (N=13) | TAC1 -> TAC4 (N=1) | TAC2 (N=9) | TAC2 -> TAC1 (N=1) | TAC2 -> TAC3 (N=1) | TAC3 (N=22) | TAC3 -> TAC1 (N=2) | TAC3 -> TAC1 -> TAC4 (N=1) | TAC3 -> TAC4 (N=2) | TAC4 (N=15) | TAC4 -> TAC1 (N=7) | TAC4 -> TAC2 (N=1) | TAC4 -> TAC3 (N=2) | Participants Enrolled But Not Treated (N=131)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 9 (15) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (3)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 6 (8) | 1 (2) | 0 (0) | 2 (2) | 4 (5) | 2 (4) | 1 (1) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 5 (13) | 0 (0) | 3 (7) | 1 (3) | 0 (0) | 9 (26) | 1 (3) | 1 (1) | 1 (6) | 10 (23) | 6 (27) | 1 (3) | 2 (9) | 2 (5)
Anorexia (Metabolism and nutrition disorders) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 9 (20) | 1 (3) | 0 (0) | 1 (2) | 3 (4) | 4 (7) | 1 (1) | 2 (4) | 1 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (8) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (8) | 1 (2) | 4 (4) | 1 (1) | 0 (0) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Corneal ulcer (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 3 (4) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 4 (11) | 1 (2) | 1 (4) | 1 (1) | 2 (3) | 4 (13) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 1 (4) | 2 (2) | 0 (0) | 1 (1) | 11 (16) | 2 (4) | 1 (1) | 2 (4) | 7 (10) | 6 (10) | 1 (1) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 1 (4) | 1 (1) | 1 (2) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 5 (9) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (2) | 0 (0) | 4 (6) | 1 (1) | 0 (0) | 7 (12) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Edema trunk (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Eye disorders - Other, Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, Peripheral shadow (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 8 (11) | 1 (4) | 4 (4) | 0 (0) | 1 (1) | 10 (16) | 1 (1) | 1 (2) | 2 (4) | 9 (12) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, Edema Limbs (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, GERD (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, Hand and Foot Syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, cellulitis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, cellulitits (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, cellutitis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, neutrophilic dermatoses (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, neutrophilic dermatosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 1 (2) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (14) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 8 (8) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 5 (13) | 2 (10) | 1 (1) | 1 (1) | 1 (2) | 2 (9) | 0 (0) | 1 (2) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (8) | 0 (0) | 3 (9) | 1 (3) | 0 (0) | 12 (27) | 1 (3) | 0 (0) | 1 (5) | 4 (6) | 2 (9) | 1 (1) | 2 (6) | 1 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 1 (4) | 4 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 1 (1) | 1 (9) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0) | 1 (2) | 1 (5) | 0 (0) | 7 (10) | 1 (1) | 0 (0) | 1 (2) | 5 (6) | 3 (7) | 0 (0) | 1 (4) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 3 (9) | 0 (0) | 2 (3) | 1 (4) | 0 (0) | 5 (10) | 1 (2) | 0 (0) | 1 (4) | 4 (6) | 3 (11) | 0 (0) | 2 (11) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (6) | 1 (1) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 1 (5) | 5 (7) | 2 (2) | 1 (1) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, TSH Inc (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 6 (11) | 0 (0) | 4 (7) | 1 (4) | 0 (0) | 4 (7) | 1 (3) | 0 (0) | 1 (7) | 3 (5) | 3 (6) | 1 (5) | 1 (10) | 1 (1)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Bilateral Arm Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Other, cramping in legs (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, muscle cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, right shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (14) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 11 (14) | 0 (0) | 1 (1) | 2 (3) | 11 (20) | 5 (10) | 0 (0) | 2 (2) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Neoplasms benign; cystic mass, tumor bleeding
Nervous system disorders - Other, vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, Vasomotor Instability (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (10) | 3 (10) | 1 (3) | 1 (2) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Pain in extremity (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 8 (11) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 5 (12) | 1 (2) | 0 (0) | 1 (2) | 11 (25) | 7 (22) | 1 (7) | 2 (9) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Psychiatric disorders - Other, labile mood; TMZ (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 8 (12) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 10 (11) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, rectal pressure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Bleeding in Plueral Fluid (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, viral illness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 3 (5) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, ingrown toe nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, lip sore & paronychia cuticles (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, hemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, pruritic rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, rash-protuberant (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, redness of left hand (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, redness, left hand (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, redness,left hand (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, skin cracking (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, skin pallor (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (15) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 6 (11) | 1 (1) | 1 (1) | 2 (3) | 8 (9) | 4 (10) | 1 (1) | 0 (0) | 1 (1)
Vulval infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 3 (7) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 7 (15) | 3 (8) | 1 (4) | 1 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/84/NCT01827384/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/84/NCT01827384/ICF_001.pdf